## CLINICAL RESEARCH DOCUMENT - COVER PAGE

| Official Study Title | Comparison of the Effects of Vaginal Cuff<br>Closure Techniques on Vaginal Length and<br>Sexual Function in Laparoscopic |
|---|---|
| | Hysterectomy |
| Document Date | 01/05/2022 |

## STUDY PROTOCOL

Patients who underwent laparoscopic hysterectomy at the Obstetrics and Gynecology Department of Abant İzzet Baysal University's Faculty of Medicine will be included in this study. During total laparoscopic hysterectomy, patients will be divided into two groups: those who underwent laparoscopic and vaginal cuff closure, based on the techniques used. Patients were recorded and evaluated based on their age, gender, parity, body mass index, complaints at presentation to our clinic, ultrasonography findings, probe curettage results, smear results, surgical indications, current chronic diseases, and previous surgical history.

The sample size was determined using a repeated-measures ANOVA test using the G\*Power 3.1.9.4 program. Accordingly, the minimum sample size to be included with a medium effect size (f=0.20), 80% statistical power, and a significance level of 0.05 was determined to be 52. To protect the study from potential losses during follow-up, an additional 10% was used to calculate 30 participants in each patient group.

Demographic data and preoperative vaginal lengths were recorded during the preoperative period. Three months after the hysterectomy, vaginal lengths were measured, and sexual life and urogenital function were evaluated. Vaginal lengths were measured without anesthesia, using the C point used for POP-Q measurement as an example. Under abdominal ultrasound control, a 5-12 mHz linear probe was used. A rigid Hegar bougie was inserted into the vagina, extending the Hegar bougie as far as it would go, marking the area externally, and measuring the length of the penis up to the hymen caruncle. This measurement was recorded as the posthysterectomy vaginal length. The Arizona Sexual Experiences Scale is a 6-point Likert-type scale consisting of 5 questions. The lowest possible score is 5, and the highest is 30. Scores of 11 or more are considered sexual dysfunction.

## STATISTICAL METHODS

Data obtained in the study will be analyzed using SPSS. Patients will be divided into two groups: laparoscopic and vaginal cuff closures, based on the techniques used during total laparoscopic hysterectomy. Power Analysis will be conducted using G Power 3.1.9.4. Statistical analyses will utilize descriptive statistics such as number, percentage, standard deviation, mean, and min/max. Student's t-test and partial correlation will be used if the data are normally distributed. The chisquare test will be used to evaluate categorical data. If the data are not normally distributed, the Mann-Whitnet U test will be used. A p<0.05 level of significance will be considered. Statistical tests will be performed using a statistical program or programs compatible with Windows.